CLINICAL TRIAL: NCT04182009
Title: A Comparison of Two Nebulisers for Performing Sputum Induction to Assess Airway Inflammation
Brief Title: A Comparison of Two Nebulisers for Sputum Induction
Acronym: FLAME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18010
Record Dates: First submitted 2019-06-12; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-06

CONDITIONS: Asthma; COPD
Keywords: Asthma; COPD; Nebuliser; Sputum Induction; Safety; Tolerability; Quality; Quantity; Physiotherapy
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omron (Other): Omron group will undergo sputum induction with the Omron nebuliser at Visit 1, followed by the Akita Jet nebuliser at Visit 2.
  Interventions: Device: Omron NE-U17 Ultrasonic nebuliser; Device: Akita Jet Inhalation System
- Akita (Active Comparator): Akita group will undergo sputum induction with the Akita Jet nebuliser at Visit 1, followed by the Omron nebuliser at Visit 2.
  Interventions: Device: Omron NE-U17 Ultrasonic nebuliser; Device: Akita Jet Inhalation System

INTERVENTIONS:
Device: Omron NE-U17 Ultrasonic nebuliser — The Omron Ultrasonic nebuliser dispenses sterile saline from a medication cup as an aerosol, which is inhaled.
Device: Akita Jet Inhalation System — The Akita Jet Inhalation System is a breath actuated nebuliser, which works with a positive pressure.

SUMMARY:
Sputum induction is considered a relatively non-invasive, reliable procedure, which can be utilised to characterise the inflammatory profile of the airways.

However, the procedure can be slightly uncomfortable for patients. This study aims to assess the differences in participants' tolerability of sputum induction, by comparing two different nebulisers when performing the procedure.

DETAILED DESCRIPTION:
This is a single centre, crossover study to compare the use of two nebulisers in the sputum induction procedure. 54 participants with stable asthma or COPD will be recruited and will attend 2 visits, at least 48 hours apart. Differences in the quality and quantity of samples and the time taken to produce a sample will be described. The main purpose is to explore the optimum device to perform the procedure, whilst protecting the safety of participants and maximising their comfort.

If participants are unable to produce a sputum sample after completion of the induction procedure, physiotherapy techniques may be performed. This is an exploratory objective to establish whether these techniques may help in the event of unsuccessful procedures.

ELIGIBILITY:
Inclusion Criteria:

* Have an ability to provide fully informed consent.
* Have a diagnosis of asthma or COPD.
* Male or female.
* Age between 18 to 75 years.

Exclusion Criteria:

* Have a post bronchodilator Forced Expiratory Volume in the first second of less than 1 litre or less than 50 percent of the predicted value.
* Have an exacerbation of asthma or COPD within the 30 days prior to the first visit.
* Have a history or current evidence of an upper or lower respiratory infection, within the 30 days prior to the first visit.
* Have any other clinically significant medical disease or uncontrolled concomitant disease, that is likely, in the opinion of the investigators to impact on the ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The tolerability to sputum induction test | During the visit, after each cycle of nebulisation (each 5 minutes)
  Checking discomfort degree due to inhalation of hypertonic saline assessed by a visual analogue scale (0 to 10)

SECONDARY OUTCOMES:
Spirometry | During the visit, up to 4 hours
  Measurement of lung function (FEV1 and FEV1%pred)
Borg Scale | During the visit, up to 4 hours
  Measurement of dyspnoea levels
The quality of sputum samples | During the processing time, 2 hours
  The analysis of squamous contamination in the sample (if >40%), viability (>65% of life cells) and quality of slide for differential cells count
The quantity of sputum samples | During the visit, up to 4 hours
  How much sputum sample was produced of sufficient quality for processing
Time to produce sample | During the visit, up to 30 minutes
  The time in minutes required to produce a sputum sample sufficient for processing
Saline quantity | During the visit, up to 30 minutes
  The amount of sterile saline required to produce a sputum sample sufficient for processing
Influence of Physiotherapy techniques | During the study visit, up to 5 minutes
  The influence of manual vibrations and Huff cough in producing a sputum sample after unsuccessful induction attempts

CONTACTS AND LOCATIONS:
Overall Officials: Professor Tim W Harrison, MBBS, BSc, MD, MSc, Principal Investigator — Professor and Honorary Consultant, University of Nottingham
Locations (1):
- Nottingham Respiratory Research Unit, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No